CLINICAL TRIAL: NCT03538041
Title: A Phase 2, Open-Label Study of INCB050465 in Participants With Autoimmune Hemolytic Anemia
Brief Title: A Study of INCB050465 in Participants With Autoimmune Hemolytic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-206; Parsaclisib (Other: Incyte Corporation); 2017-003652-22 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Hemolytic Anemia
Keywords: autoimmune hemolytic anemia; phosphatidylinositol 3-kinase (PI3K) inhibitor
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Hereditary Sensory and Autonomic Neuropathies | interventions — parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parsaclisib 1 mg QD (Experimental): Parsaclisib at 1 milligram (mg) once daily (QD) for 12 weeks followed by extension period, with a dose-increase option (to 2.5 mg QD) at Week 6 for participants who fulfill dose increase criteria.
  Interventions: Drug: Parsaclisib
- Parsaclisib 2.5 mg QD (Experimental): Parsaclisib at 2.5 mg QD for 12 weeks followed by extension period.
  Interventions: Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Parsaclisib administered orally.
  Other Names: INCB050465

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of parsaclisib administered orally to participants with autoimmune hemolytic anemia (AIHA) who have decreased hemoglobin and evidence of ongoing hemolysis that requires treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIHA based on the presence of hemolytic anemia and serological evidence of anti-erythrocyte antibodies, detectable by the direct antiglobulin test.
* Participants who have disease progression after treatment with standard therapies that are known to confer clinical benefit, or who are intolerant to treatment, or who refuse standard treatment. There is no limit to the number of prior treatment regimens.
* Hemoglobin 7 to 10 g/dL.
* No evidence of a lymphoproliferative malignancy or other autoimmune-related underlying conditions.
* Eastern Cooperative Oncology Group performance status of 0 to 2.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Concurrent conditions and history of other protocol-specified diseases.
* ANC < 1.5 × 10^9/L.
* Platelet count < 100 × 10^9/L.
* Severely impaired liver function.
* Impaired renal function with estimated creatinine clearance less than 45 mL/min.
* Anti-phospholipid antibodies positive or elevated anti-streptolysin antibodies.
* Positive serology test results for hepatitis B surface antigen or core antibody, or hepatitis C virus antibody with detectable RNA at screening, consistent with active or chronic infection.
* Known HIV infection or positivity on immunoassay.
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically meaningful.
* Known hypersensitivity or severe reaction to parsaclisib or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Butler, MD, Study Director — Incyte Corporation
Locations (12):
- United States (6):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Health System Inc., Dba the University of Tn Medical Center, Knoxville, Tennessee
- Allgemeines Krankenhaus Der Stadt Wien, Vienna, Austria
- France (2):
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier Regional Universitaire (Chru) de Lille, Lille
- Italy (3):
  - Fondazione Irccs Ca Granda Ospedale Maggiore, Milan
  - UNIVERSITï¿½ DI NAPOLI FEDERICO II, Napoli
  - AZIENDA OSPEDALIERO UNIVERSITARIA MAGGIORE DELLA CARITï¿½ DI NOVARA, Novara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barcellini W, Pane F, Patriarca A, Murakhovskaya I, Terriou L, DeSancho MT, Hanna WT, Leopold L, Rappold E, Szeto K, Wei S, Jager U. Parsaclisib for the treatment of primary autoimmune hemolytic anemia: Results from a phase 2, open-label study. Am J Hematol. 2024 Dec;99(12):2313-2320. doi: 10.1002/ajh.27493. Epub 2024 Oct 22. PMID 39435908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 25 participants enrolled in 8 sites in Austria, France, Italy, and the United States.
Groups:
- Parsaclisib 1 mg QD: Participants received oral parsaclisib once daily (QD) for 12 weeks. Participants initially received parsaclisib 1 milligram (mg) QD. At Week 6, participants who continued to require transfusions or did not attain a meaningful clinical response (at least a stabilization of a ≥ 2 grams per deciliter [g/dL] increase in hemoglobin from Baseline to Week 6) may have had their dose increased, with sponsor preapproval, to parsaclisib 2.5 mg QD until Week 12. If there were any tolerability issues in individual participants who received 2.5 mg, the dose could have been decreased to 1 mg. Participants who continued to receive clinical benefit after the 12-week Treatment Period could have entered into an Extension Period, during which they, with sponsor approval, continued to receive parsaclisib 1 mg QD or 2.5 mg QD until the drug was available through another clinical study, or was commercially available, or the sponsor stopped the study or the study drug development. Following the last dose of parsaclisib, in either the Treatment Period (for participants not entering the Extension Period) or the Extension Period, participants were eligible for a 12-week (3-month) follow-up period.
- Parsaclisib 2.5 mg QD: Participants received oral parsaclisib 2.5 mg QD for 12 weeks. If there were any tolerability issues in individual participants, the dose could have been decreased to 1 mg. Participants who continued to receive clinical benefit after the 12-week Treatment Period could have entered into an Extension Period, during which they, with sponsor approval, continued to receive parsaclisib 2.5 mg QD until the drug was available through another clinical study, or was commercially available, or the sponsor stopped the study or the study drug development. Following the last dose of parsaclisib, in either the Treatment Period (for participants not entering the Extension Period) or the Extension Period, participants were eligible for a 12-week (3-month) follow-up period.
Period: 12-Week Treatment Period
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Started | 10 | 15
Completed | 9 | 13
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Extension Period
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Started | 7 (These participants completed the 24-week Treatment Period and were eligible for an extension of treatment based on their clinical response.) | 11 (These participants completed the 24-week Treatment Period and were eligible for an extension of treatment based on their clinical response.)
Completed | 0 | 0
Not Completed | 7 | 11
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Lack of Efficacy | 1 | 4
Not completed — Transitioned to Rollover Study | 1 | 4
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD | Total
Number analyzed (Participants) | 10 | 15 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (9.63) | 60.3 (20.74) | 61.6 (16.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 14 | 23
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 9 | 14 | 23
  Black/African-American | 1 | 0 | 1
  Captured as "Other" | 0 | 1 | 1
Hemoglobin [Mean (Standard Deviation); unit: grams per deciliter (g/dL)] | 9.1 (0.80) | 8.7 (0.85) | 8.9 (0.83)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Attaining a Complete Response at Any Visit From Week 6 to Week 12
Description: A complete response was defined as hemoglobin >12 grams per deciliter (g/dL) not attributed to a transfusion effect and the normalization of hemolytic markers. No transfusion effect was defined as > 1 week since the last transfusion.
Time Frame: Week 6 to Week 12
Population: Full Analysis Set: all participants who enrolled in the study who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants | 20.0 | 40.0

2. Primary Outcome: Percentage of Participants Attaining a Partial Response at Any Visit From Week 6 to Week 12
Description: A partial response was defined as hemoglobin 10-12 g/dL or at least a 2 g/dL increase from Baseline not attributed to a transfusion effect and the normalization of hemolytic markers. No transfusion effect was defined as > 1 week since the last transfusion.
Time Frame: Week 6 to Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants | 60.0 | 66.7

3. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy, or required changes in the study drug. Anemia and transfusions should not have been reported as AEs unless they represented a clinically meaningful decrease from Baseline in hemoglobin. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to 1638 days
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
Participants | 10 | 15

4. Secondary Outcome: Percentage of Participants Attaining a Complete Response During Post-Baseline Visits
Description: A complete response was defined as hemoglobin >12 g/dL) not attributed to a transfusion effect and the normalization of hemolytic markers. No transfusion effect was defined as > 1 week since the last transfusion.
Time Frame: up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants
  Week 1 | 0.0 | 6.7
  Week 2 | 10.0 | 6.7
  Week 4: number analyzed (Participants) | 9 | 14
  Week 4 | 22.2 | 21.4
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 22.2 | 28.6
  Week 8: number analyzed (Participants) | 9 | 13
  Week 8 | 22.2 | 23.1
  Week 10: number analyzed (Participants) | 9 | 13
  Week 10 | 22.2 | 23.1
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 22.2 | 42.9
  Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Follow-up Month 1 | 0.0 | 0.0
  Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Follow-up Month 2 | 0.0 | 0.0
  Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Follow-up Month 3 | 0.0 | 0.0
  Extension End of Treatment: number analyzed (Participants) | 6 | 10
  Extension End of Treatment | 50.0 | 50.0

5. Secondary Outcome: Percentage of Participants Attaining a Partial Response During Post-Baseline Visits
Description: as for outcome 2
Time Frame: up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants
  Week 1 | 50.0 | 53.3
  Week 2 | 50.0 | 66.7
  Week 4: number analyzed (Participants) | 9 | 14
  Week 4 | 44.4 | 64.3
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 44.4 | 50.0
  Week 8: number analyzed (Participants) | 9 | 13
  Week 8 | 55.6 | 61.5
  Week 10: number analyzed (Participants) | 9 | 13
  Week 10 | 55.6 | 61.5
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 55.6 | 64.3
  Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Follow-up Month 1 | 50.0 | 0.0
  Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Follow-up Month 2 | 0.0 | 0.0
  Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Follow-up Month 3 | 0.0 | 50.0
  Extension End of Treatment: number analyzed (Participants) | 6 | 10
  Extension End of Treatment | 83.3 | 50.0

6. Secondary Outcome: Percentage of Participants Attaining a ≥ 2 g/dL Increase in Hemoglobin From Baseline
Description: Hemoglobin levels were assessed throughout the study.
Time Frame: up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants
  Week 1 | 0.0 | 26.7
  Week 2 | 10.0 | 46.7
  Week 4: number analyzed (Participants) | 9 | 14
  Week 4 | 22.2 | 42.9
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 22.2 | 35.7
  Week 8: number analyzed (Participants) | 9 | 13
  Week 8 | 33.3 | 38.5
  Week 10: number analyzed (Participants) | 9 | 13
  Week 10 | 22.2 | 46.2
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 33.3 | 50.0
  Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Follow-up Month 1 | 0.0 | 0.0
  Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Follow-up Month 2 | 0.0 | 0.0
  Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Follow-up Month 3 | 0.0 | 0.0
  Extension End of Treatment: number analyzed (Participants) | 6 | 10
  Extension End of Treatment | 66.7 | 50.0

7. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
grams per deciliter (g/dL)
  Baseline | 9.1 (0.80) | 8.7 (0.85)
  Change from Baseline at Week 1 | 0.9 (0.84) | 1.2 (1.30)
  Change from Baseline at Week 2 | 0.6 (0.96) | 1.5 (1.75)
  Change from Baseline at Week 4: number analyzed (Participants) | 9 | 14
  Change from Baseline at Week 4 | 0.9 (1.06) | 1.6 (1.79)
  Change from Baseline at Week 6: number analyzed (Participants) | 9 | 14
  Change from Baseline at Week 6 | 1.2 (0.80) | 1.7 (1.96)
  Change from Baseline at Week 8: number analyzed (Participants) | 9 | 13
  Change from Baseline at Week 8 | 1.2 (1.14) | 2.0 (2.07)
  Change from Baseline at Week 10: number analyzed (Participants) | 9 | 13
  Change from Baseline at Week 10 | 1.3 (1.14) | 2.1 (2.22)
  Change from Baseline at Week 12: number analyzed (Participants) | 9 | 14
  Change from Baseline at Week 12 | 1.3 (1.46) | 2.5 (2.67)
  Change from Baseline at Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Change from Baseline at Follow-up Month 1 | 0.1 (1.06) | -0.4 (0.72)
  Change from Baseline at Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Change from Baseline at Follow-up Month 2 | -0.1 (0.28) | -0.2 (0.28)
  Change from Baseline at Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Change from Baseline at Follow-up Month 3 | 0.5 (0.92) | 0.2 (1.63)
  Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 6 | 10
  Change from Baseline at Extension End of Treatment | 2.8 (2.70) | 2.6 (2.73)

8. Secondary Outcome: Percentage Change From Baseline in Hemoglobin
Description: Percentage change from Baseline was calculated as: ([post-Baseline value minus the Baseline value] / Baseline value) x 100.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percent change
  Week 1 | 10.1 (9.23) | 14.4 (16.31)
  Week 2 | 6.0 (10.26) | 18.5 (20.71)
  Week 4: number analyzed (Participants) | 9 | 14
  Week 4 | 9.9 (10.83) | 19.2 (20.65)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 13.3 (8.35) | 19.5 (22.35)
  Week 8: number analyzed (Participants) | 9 | 13
  Week 8 | 12.7 (12.16) | 23.4 (24.57)
  Week 10: number analyzed (Participants) | 9 | 13
  Week 10 | 14.1 (11.54) | 25.1 (26.30)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 13.9 (15.72) | 30.2 (33.95)
  Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Follow-up Month 1 | 0.0 (12.26) | -4.1 (7.92)
  Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Follow-up Month 2 | -1.0 (3.18) | -2.0 (2.89)
  Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Follow-up Month 3 | 5.7 (11.14) | 2.0 (17.32)
  Extension End of Treatment: number analyzed (Participants) | 6 | 10
  Extension End of Treatment | 31.6 (33.86) | 30.9 (33.52)

9. Secondary Outcome: Percentage of Participants Requiring Transfusions
Description: A participant was defined to have required a transfusion if his or her last transfusion was within 7 days of the visit date.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants
  Week 1 | 0.0 | 6.7
  Week 2 | 0.0 | 0.0
  Week 4: number analyzed (Participants) | 9 | 14
  Week 4 | 22.2 | 0.0
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 0.0 | 0.0
  Week 8: number analyzed (Participants) | 9 | 13
  Week 8 | 0.0 | 15.4
  Week 10: number analyzed (Participants) | 9 | 13
  Week 10 | 0.0 | 7.7
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 0.0 | 0.0
  Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Follow-up Month 1 | 0.0 | 0.0
  Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Follow-up Month 2 | 0.0 | 0.0
  Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Follow-up Month 3 | 0.0 | 0.0
  Extension End of Treatment: number analyzed (Participants) | 6 | 10
  Extension End of Treatment | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants Who Achieved Normalization of Hemoglobin, Haptoglobin, Lactate Dehydrogenase (LDH), Reticulocyte Count, Total Bilirubin, Direct Bilirubin, and Indirect Bilirubin
Description: Normalization was determined by the Investigator based on normal ranges for the clinical reference laboratory.
Time Frame: up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants
  Hemoglobin, Week 1 | 0.0 | 6.7
  Hemoglobin, Week 2 | 0.0 | 6.7
  Hemoglobin, Week 4: number analyzed (Participants) | 9 | 14
  Hemoglobin, Week 4 | 0.0 | 14.3
  Hemoglobin, Week 6: number analyzed (Participants) | 9 | 14
  Hemoglobin, Week 6 | 0.0 | 21.4
  Hemoglobin, Week 8: number analyzed (Participants) | 9 | 13
  Hemoglobin, Week 8 | 0.0 | 15.4
  Hemoglobin, Week 10: number analyzed (Participants) | 9 | 13
  Hemoglobin, Week 10 | 0.0 | 15.4
  Hemoglobin, Week 12: number analyzed (Participants) | 9 | 14
  Hemoglobin, Week 12 | 11.1 | 35.7
  Hemoglobin, Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Hemoglobin, Follow-up Month 1 | 0.0 | 0.0
  Hemoglobin, Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Hemoglobin, Follow-up Month 2 | 0.0 | 0.0
  Hemoglobin, Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Hemoglobin, Follow-up Month 3 | 0.0 | 0.0
  Haptoglobin, Week 1: number analyzed (Participants) | 8 | 9
  Haptoglobin, Week 1 | 12.5 | 22.2
  Haptoglobin, Week 2: number analyzed (Participants) | 6 | 11
  Haptoglobin, Week 2 | 0.0 | 18.2
  Haptoglobin, Week 4: number analyzed (Participants) | 7 | 13
  Haptoglobin, Week 4 | 14.3 | 15.4
  Haptoglobin, Week 6: number analyzed (Participants) | 7 | 13
  Haptoglobin, Week 6 | 14.3 | 23.1
  Haptoglobin, Week 8: number analyzed (Participants) | 7 | 9
  Haptoglobin, Week 8 | 0.0 | 11.1
  Haptoglobin, Week 10: number analyzed (Participants) | 8 | 7
  Haptoglobin, Week 10 | 12.5 | 14.3
  Haptoglobin, Week 12: number analyzed (Participants) | 7 | 12
  Haptoglobin, Week 12 | 14.3 | 25.0
  Haptoglobin, Follow-up Month 2: number analyzed (Participants) | 1 | 0
  Haptoglobin, Follow-up Month 2 | 0.0 |
  LDH, Week 1: number analyzed (Participants) | 8 | 10
  LDH, Week 1 | 12.5 | 10.0
  LDH, Week 2: number analyzed (Participants) | 9 | 12
  LDH, Week 2 | 11.1 | 16.7
  LDH, Week 4: number analyzed (Participants) | 8 | 14
  LDH, Week 4 | 12.5 | 21.4
  LDH, Week 6: number analyzed (Participants) | 7 | 14
  LDH, Week 6 | 14.3 | 14.3
  LDH, Week 8: number analyzed (Participants) | 8 | 11
  LDH, Week 8 | 25.0 | 9.1
  LDH, Week 10 | 33.3 | 9.1
  LDH, Week 12: number analyzed (Participants) | 8 | 13
  LDH, Week 12 | 25.0 | 15.4
  LDH, Follow-up Month 2: number analyzed (Participants) | 1 | 0
  LDH, Follow-up Month 2 | 0.0 |
  Reticulocytes, Week 1: number analyzed (Participants) | 10 | 14
  Reticulocytes, Week 1 | 20.0 | 14.3
  Reticulocytes, Week 2: number analyzed (Participants) | 7 | 15
  Reticulocytes, Week 2 | 28.6 | 20.0
  Reticulocytes, Week 4: number analyzed (Participants) | 8 | 14
  Reticulocytes, Week 4 | 25.0 | 28.6
  Reticulocytes, Week 6: number analyzed (Participants) | 9 | 14
  Reticulocytes, Week 6 | 22.2 | 28.6
  Reticulocytes, Week 8: number analyzed (Participants) | 8 | 12
  Reticulocytes, Week 8 | 25.0 | 25.0
  Reticulocytes, Week 10: number analyzed (Participants) | 6 | 12
  Reticulocytes, Week 10 | 33.3 | 25.0
  Reticulocytes, Week 12: number analyzed (Participants) | 8 | 13
  Reticulocytes, Week 12 | 37.5 | 23.1
  Reticulocytes, Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Reticulocytes, Follow-up Month 1 | 50.0 | 0.0
  Reticulocytes, Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Reticulocytes, Follow-up Month 2 | 50.0 | 0.0
  Reticulocytes, Follow-up Month 3: number analyzed (Participants) | 2 | 1
  Reticulocytes, Follow-up Month 3 | 50.0 | 0.0
  Total bilirubin, Week 1 | 30.0 | 40.0
  Total bilirubin, Week 2 | 20.0 | 40.0
  Total bilirubin, Week 4: number analyzed (Participants) | 9 | 14
  Total bilirubin, Week 4 | 33.3 | 42.9
  Total bilirubin, Week 6: number analyzed (Participants) | 9 | 14
  Total bilirubin, Week 6 | 33.3 | 42.9
  Total bilirubin, Week 8: number analyzed (Participants) | 9 | 12
  Total bilirubin, Week 8 | 44.4 | 50.0
  Total bilirubin, Week 10: number analyzed (Participants) | 9 | 11
  Total bilirubin, Week 10 | 44.4 | 36.4
  Total bilirubin, Week 12: number analyzed (Participants) | 9 | 14
  Total bilirubin, Week 12 | 44.4 | 50.0
  Total bilirubin, Follow-up Month 2: number analyzed (Participants) | 1 | 0
  Total bilirubin, Follow-up Month 2 | 100.0 |
  Direct bilirubin, Week 1: number analyzed (Participants) | 6 | 8
  Direct bilirubin, Week 1 | 0.0 | 25.0
  Direct bilirubin, Week 2: number analyzed (Participants) | 8 | 9
  Direct bilirubin, Week 2 | 12.5 | 22.2
  Direct bilirubin, Week 4: number analyzed (Participants) | 6 | 8
  Direct bilirubin, Week 4 | 0.0 | 12.5
  Direct bilirubin, Week 6: number analyzed (Participants) | 6 | 8
  Direct bilirubin, Week 6 | 0.0 | 25.0
  Direct bilirubin, Week 8: number analyzed (Participants) | 5 | 5
  Direct bilirubin, Week 8 | 0.0 | 20.0
  Direct bilirubin, Week 10: number analyzed (Participants) | 5 | 7
  Direct bilirubin, Week 10 | 0.0 | 14.3
  Direct bilirubin, Week 12: number analyzed (Participants) | 5 | 7
  Direct bilirubin, Week 12 | 0.0 | 28.6
  Indirect bilirubin, Week 1: number analyzed (Participants) | 6 | 8
  Indirect bilirubin, Week 1 | 0.0 | 12.5
  Indirect bilirubin, Week 2: number analyzed (Participants) | 8 | 9
  Indirect bilirubin, Week 2 | 0.0 | 0.0
  Indirect bilirubin, Week 4: number analyzed (Participants) | 6 | 8
  Indirect bilirubin, Week 4 | 0.0 | 0.0
  Indirect bilirubin, Week 6: number analyzed (Participants) | 6 | 8
  Indirect bilirubin, Week 6 | 0.0 | 0.0
  Indirect bilirubin, Week 8: number analyzed (Participants) | 5 | 5
  Indirect bilirubin, Week 8 | 0.0 | 0.0
  Indirect bilirubin, Week 10: number analyzed (Participants) | 5 | 7
  Indirect bilirubin, Week 10 | 0.0 | 0.0
  Indirect bilirubin, Week 12: number analyzed (Participants) | 5 | 7
  Indirect bilirubin, Week 12 | 0.0 | 0.0

11. Secondary Outcome: Percentage of Participants Requiring a Prednisone Dose Change (Increase or Decrease)
Description: Prednisone use was monitored throughout the study.
Time Frame: up to 1638 days
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
percentage of participants
  Week 1, increased | 0.0 | 6.7
  Week 1, decreased | 20.0 | 6.7
  Week 2, increased | 0.0 | 0.0
  Week 2, decreased | 20.0 | 13.3
  Week 4, increased | 0.0 | 0.0
  Week 4, decreased | 10.0 | 6.7
  Week 6, increased | 0.0 | 0.0
  Week 6, decreased | 10.0 | 6.7
  Week 8, increased | 0.0 | 0.0
  Week 8, decreased | 10.0 | 6.7
  Week 10, increased | 0.0 | 0.0
  Week 10, decreased | 10.0 | 6.7
  Week 12, increased | 0.0 | 0.0
  Week 12, decreased | 10.0 | 20.0
  Extension End of Treatment, increased | 10.0 | 6.7
  Extension End of Treatment, decreased | 10.0 | 6.7

12. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Subscale Scores
Description: The FACIT-F subscale is a 13-item instrument designed to assess fatigue/tiredness and its impact on daily activities and functioning in a number of chronic diseases. Participants were asked to respond to 13 statements that people with the illness have said are important on the following scale: 0, not at all; 1, a little bit; 2, somewhat; 3, quite a bit; 4, very much. Participants were asked to indicate the response as it applied to the last 7 days. The total fatigue subscale score ranges from 0 to 52; a higher score indicates more severe impact on daily activities and functioning.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
scores on a scale
  Baseline | 32.6 (12.80) | 30.1 (13.88)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 6.7 (12.44) | 8.2 (9.28)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 6.2 (16.08) | 5.4 (15.49)
  Follow-up Month 1: number analyzed (Participants) | 2 | 3
  Follow-up Month 1 | 2.0 (2.83) | 2.3 (10.69)
  Follow-up Month 2: number analyzed (Participants) | 2 | 2
  Follow-up Month 2 | 1.5 (7.78) | 7.0 (15.56)
  Follow-up Month 3: number analyzed (Participants) | 2 | 2
  Follow-up Month 3 | -2.0 (21.21) | 13.0 (14.14)

13. Secondary Outcome: Mean Cmax of Parsaclisib
Description: Cmax was defined as the maximum observed concentration. Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: Pharmacokinetic (PK)/Pharmacodynamic (PD) Evaluable Population: all participants who received at least 1 dose of study drug and provided at least 1 postdose blood sample for PK or biomarker assessment. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per Liter (nmol/L)
Groups:
- Cohort 1: Parsaclisib 1 mg QD: Participants who received oral parsaclisib 1 mg QD for 12 weeks and did not qualify for a dose increase to 2.5 mg QD starting at Week 6 (they did not continue to require transfusions or they attained a meaningful clinical response [at least a stabilization of a ≥ 2 g/dL increase in hemoglobin from Baseline to Week 6]).
- Cohort 1: Parsaclisib 2.5 mg QD: Participants who initially received oral parsaclisib 1 mg QD, but had their dose increased, with sponsor preapproval, to 2.5 mg QD starting at Week 6 (up to Week 12) because they continued to require transfusions or did not attain a meaningful clinical response (at least a stabilization of a ≥ 2 g/dL increase in hemoglobin from Baseline to Week 6).
- Cohort 2: Parsaclisib 2.5 mg QD: Participants received oral parsaclisib 2.5 mg QD for 12 weeks.
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
nanomoles per Liter (nmol/L)
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 94.9 (33.5) |  | 191 (56.2)
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 107 (17.8) | 219 (45.2) | 199 (39.7)
Statistical Analysis 1: Comparison: Cohort 1: Parsaclisib 1 mg QD vs Cohort 2: Parsaclisib 2.5 mg QD; Week 2; Test type: Superiority; p = 0.2815, ANOVA

14. Secondary Outcome: Mean Tmax of Parsaclisib
Description: tmax was defined as the time to the maximum concentration. Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: PK/PD Evaluable Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
hours
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 1.00 [0.00 to 2.07] |  | 1.00 [0.00 to 3.33]
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 1.00 [1.00 to 1.05] | 1.04 [0.917 to 2.00] | 1.02 [0.833 to 4.00]
Statistical Analysis 1: Comparison: Cohort 1: Parsaclisib 1 mg QD vs Cohort 2: Parsaclisib 2.5 mg QD; Week 2; Test type: Superiority; p = 0.2921, Kruskal-Wallis

15. Secondary Outcome: Mean Cmin of Parsaclisib
Description: Cmin was defined as the minimum observed concentration over the dose interval. Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: PK/PD Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
nmol/L
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 20.0 (88.7) |  | 32.3 (55.4)
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 14.2 (80.9) | 39.4 (26.1) | 25.5 (91.4)
Statistical Analysis 1: Comparison: Cohort 1: Parsaclisib 1 mg QD vs Cohort 2: Parsaclisib 2.5 mg QD; Week 2; Test type: Superiority; p = 0.1267, ANOVA

16. Secondary Outcome: Mean AUC0-4 of Parsaclisib
Description: AUC0-4 was defined as the area under the concentration-time curve from time = 0 to 4 hours postdose. Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: PK/PD Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nmol/L
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
hours*nmol/L
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 260 (24.0) |  | 542 (46.7)
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 287 (5.73) | 631 (41.9) | 524 (50.8)
Statistical Analysis 1: Comparison: Cohort 1: Parsaclisib 1 mg QD vs Cohort 2: Parsaclisib 2.5 mg QD; Week 2; Test type: Superiority; p = 0.2676, ANOVA

17. Secondary Outcome: Mean AUC0-t of Parsaclisib
Description: AUC0-t was defined as the area under the concentration-time curve from time = 0 to the last measureable concentration at time = t. Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: PK/PD Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nmol/L
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
hours*nmol/L
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 260 (24.0) |  | 553 (41.3)
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 287 (5.73) | 633 (42.4) | 524 (50.8)

18. Secondary Outcome: Mean Clast of Parsaclisib
Description: Clast was defined as the last measurable concentration (above the quantification limit). Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: PK/PD Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
nmol/L
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 59.6 (21.3) |  | 128 (53.3)
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 62.4 (7.31) | 134 (54.2) | 138 (42.3)

19. Secondary Outcome: Mean Tlast of Parsaclisib
Description: Tlast was defined as the time of the last measurable concentration (above the quantification limit). Participants in Cohort 1 were not eligible to receive parsaclisib 2.5 mg at Week 2.
Time Frame: predose at Weeks 1 and 12; predose and 1, 2, and 4 hours postdose at Weeks 2 and 8
Population: PK/PD Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Cohort 1: Parsaclisib 1 mg QD | Cohort 1: Parsaclisib 2.5 mg QD | Cohort 2: Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 6 | 15
hours
  Week 2: number analyzed (Participants) | 9 | 0 | 15
  Week 2 | 3.85 (4.77) |  | 3.98 (9.67)
  Week 8: number analyzed (Participants) | 3 | 6 | 11
  Week 8 | 3.83 (5.84) | 3.92 (3.71) | 3.84 (6.56)

20. Secondary Outcome: Change From Baseline in Reticulocyte Count
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter (10^9 cells/L)
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
10^9 cells per Liter (10^9 cells/L)
  Baseline of the Treatment Period (TP): number analyzed (Participants) | 10 | 14
  Baseline of the Treatment Period (TP) | 240.7460 (110.0788) | 268.1429 (128.3266)
  Change from Baseline at Week 1 of the TP: number analyzed (Participants) | 10 | 13
  Change from Baseline at Week 1 of the TP | -6.8244 (75.4853) | -37.9910 (90.4026)
  Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 7 | 14
  Change from Baseline at Week 2 of the TP | -17.2571 (87.7742) | -55.4934 (88.8296)
  Change from Baseline at Week 4 of the TP: number analyzed (Participants) | 8 | 13
  Change from Baseline at Week 4 of the TP | -24.8375 (52.5381) | -67.8155 (86.6172)
  Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 9 | 13
  Change from Baseline at Week 6 of the TP | -45.4739 (61.9611) | -46.3599 (106.7383)
  Change from Baseline at Week 8 of the TP: number analyzed (Participants) | 8 | 11
  Change from Baseline at Week 8 of the TP | -43.0819 (87.7012) | -74.8763 (97.2582)
  Change from Baseline at Week 10 of the TP: number analyzed (Participants) | 6 | 11
  Change from Baseline at Week 10 of the TP | -24.3667 (55.3112) | -50.4759 (104.4132)
  Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 8 | 12
  Change from Baseline at Week 12 of the TP | -27.1250 (63.3308) | -80.7566 (112.2789)
  Change from Baseline at Follow-up Month 1 of the TP: number analyzed (Participants) | 2 | 3
  Change from Baseline at Follow-up Month 1 of the TP | 0.0000 (26.1630) | 2.6297 (16.8763)
  Change from Baseline at Follow-up Month 2 of the TP: number analyzed (Participants) | 2 | 2
  Change from Baseline at Follow-up Month 2 of the TP | -18.2000 (17.6777) | -16.4500 (23.2638)
  Change from Baseline at Follow-up Month 3 of the TP: number analyzed (Participants) | 2 | 1
  Change from Baseline at Follow-up Month 3 of the TP | -31.1500 (11.2430) | -131.900 (NA) — Standard deviation cannot be calculated for a single participant.
  Baseline of the Extension Period (EP): number analyzed (Participants) | 7 | 10
  Baseline of the Extension Period (EP) | 233.3086 (121.4996) | 243.9526 (104.4420)
  Change from Baseline at End of Treatment during the EP: number analyzed (Participants) | 5 | 9
  Change from Baseline at End of Treatment during the EP | 184.4096 (102.9469) | 191.7013 (131.3629)

21. Secondary Outcome: Change From Baseline in Cardiolipin Immunoglobulin G (IgG) Antibody and Cardiolipin Immunoglobulin M (IgM) Antibody
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 9 | 12
micrograms per milliliter (µg/mL)
  IgG at Baseline | 0.0 (0.00) | 5.8 (20.21)
  Change from Baseline in IgG at Week 12: number analyzed (Participants) | 0 | 0
  IgM at Baseline | 0.0 (0.00) | 1.7 (3.24)
  Change from Baseline in IgM at Week 12: number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Change From Baseline in Cold Hemagglutinin Levels
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: titer
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 2 | 6
titer
  Baseline | 3200 (2715.29) | 11206.67 (10309.03)
  Change from Baseline at Week 12: number analyzed (Participants) | 2 | 2
  Change from Baseline at Week 12 | -1760 (1131.371) | 960 (1357.645)

23. Secondary Outcome: Change From Baseline in Haptoglobin, Total Bilirubin, Direct Bilirubin, and Indirect Bilirubin
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles (µmol)/L
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
micromoles (µmol)/L
  Haptoglobin, Baseline of the TP: number analyzed (Participants) | 10 | 14
  Haptoglobin, Baseline of the TP | 0.00 (0.000) | 0.81 (3.020)
  Haptoglobin, Change from Baseline at Week 1 of the TP: number analyzed (Participants) | 8 | 9
  Haptoglobin, Change from Baseline at Week 1 of the TP | 0.65 (1.838) | 1.20 (1.879)
  Haptoglobin, Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 6 | 11
  Haptoglobin, Change from Baseline at Week 2 of the TP | 0.00 (0.000) | 0.90 (1.640)
  Haptoglobin, Change from Baseline at Week 4 of the TP: number analyzed (Participants) | 7 | 13
  Haptoglobin, Change from Baseline at Week 4 of the TP | 0.73 (1.928) | 0.75 (2.066)
  Haptoglobin, Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 7 | 13
  Haptoglobin, Change from Baseline at Week 6 of the TP | 1.09 (2.873) | 2.48 (5.069)
  Haptoglobin, Change from Baseline at Week 8 of the TP: number analyzed (Participants) | 7 | 9
  Haptoglobin, Change from Baseline at Week 8 of the TP | 0.00 (0.000) | 1.36 (3.293)
  Haptoglobin, Change from Baseline at Week 10 of the TP: number analyzed (Participants) | 8 | 7
  Haptoglobin, Change from Baseline at Week 10 of the TP | 1.55 (3.579) | 1.04 (2.759)
  Haptoglobin, Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 7 | 12
  Haptoglobin, Change from Baseline at Week 12 of the TP | 0.73 (1.928) | 1.34 (2.654)
  Haptoglobin, Change from Baseline at Follow-up Month 2 of the TP: number analyzed (Participants) | 1 | 0
  Haptoglobin, Change from Baseline at Follow-up Month 2 of the TP | 0.00 (NA) — Standard deviation cannot be calculated for a single participant. |
  Haptoglobin, Baseline of the EP: number analyzed (Participants) | 7 | 11
  Haptoglobin, Baseline of the EP | 0.0000 (0.0000) | 0.0000 (0.0000)
  Haptoglobin, Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 5 | 7
  Haptoglobin, Change from Baseline at Extension End of Treatment | 2.9200 (5.4906) | 4.0000 (5.2386)
  Indirect bilirubin, Baseline of the TP: number analyzed (Participants) | 6 | 14
  Indirect bilirubin, Baseline of the TP | 32.7 (13.29) | 36.1 (22.77)
  Indirect bilirubin, Change from Baseline at Week 1 of the TP: number analyzed (Participants) | 5 | 8
  Indirect bilirubin, Change from Baseline at Week 1 of the TP | -6.2 (7.66) | -11.9 (18.73)
  Indirect bilirubin, Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 6 | 9
  Indirect bilirubin, Change from Baseline at Week 2 of the TP | -2.3 (4.59) | -11.6 (17.67)
  Indirect bilirubin, Change from Baseline at Week 4 of the TP: number analyzed (Participants) | 5 | 8
  Indirect bilirubin, Change from Baseline at Week 4 of the TP | -7.6 (9.63) | -11.1 (21.63)
  Indirect bilirubin, Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 5 | 8
  Indirect bilirubin, Change from Baseline at Week 6 of the TP | -11.0 (14.20) | -13.6 (22.39)
  Indirect bilirubin, Change from Baseline at Week 8 of the TP: number analyzed (Participants) | 4 | 5
  Indirect bilirubin, Change from Baseline at Week 8 of the TP | -3.5 (15.63) | -16.8 (34.58)
  Indirect bilirubin, Change from Baseline at Week 10 of the TP: number analyzed (Participants) | 4 | 7
  Indirect bilirubin, Change from Baseline at Week 10 of the TP | -6.5 (9.95) | -14.7 (25.44)
  Indirect bilirubin, Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 4 | 7
  Indirect bilirubin, Change from Baseline at Week 12 of the TP | -2.5 (13.03) | -17.0 (24.39)
  Indirect bilirubin, Baseline of the EP: number analyzed (Participants) | 4 | 10
  Indirect bilirubin, Baseline of the EP | 35.2500 (15.7348) | 33.4000 (24.5185)
  Indirect bilirubin, Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 1 | 3
  Indirect bilirubin, Change from Baseline at Extension End of Treatment | -34.3610 (NA) — Standard deviation cannot be calculated for a single participant. | -0.7057 (8.3763)
  Total bilirubin, Baseline of the TP | 34.7 (19.58) | 54.3 (51.65)
  Total bilirubin, Change from Baseline at Week 1 of the TP | -2.8 (14.65) | -18.3 (34.92)
  Total bilirubin, Change from Baseline at Week 2 of the TP | 1.7 (11.94) | -18.7 (34.44)
  Total bilirubin, Change from Baseline at Week 4 of the TP: number analyzed (Participants) | 9 | 14
  Total bilirubin, Change from Baseline at Week 4 of the TP | -2.2 (16.53) | -19.5 (35.14)
  Total bilirubin, Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 9 | 14
  Total bilirubin, Change from Baseline at Week 6 of the TP | -3.6 (22.82) | -21.6 (31.27)
  Total bilirubin, Change from Baseline at Week 8 of the TP: number analyzed (Participants) | 9 | 12
  Total bilirubin, Change from Baseline at Week 8 of the TP | -0.9 (17.24) | -22.3 (41.89)
  Total bilirubin, Change from Baseline at Week 10 of the TP: number analyzed (Participants) | 9 | 11
  Total bilirubin, Change from Baseline at Week 10 of the TP | -2.7 (17.59) | -23.6 (29.83)
  Total bilirubin, Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 9 | 14
  Total bilirubin, Change from Baseline at Week 12 of the TP | -2.0 (14.86) | -21.3 (24.03)
  Total bilirubin, Change from Baseline at Follow-up Month 2 of the TP: number analyzed (Participants) | 1 | 0
  Total bilirubin, Change from Baseline at Follow-up Month 2 of the TP | 2.0 (NA) — Standard deviation cannot be calculated for a single participant. |
  Total bilirubin, Baseline of the EP: number analyzed (Participants) | 7 | 11
  Total bilirubin, Baseline of the EP | 34.7143 (22.2165) | 40.0000 (27.6586)
  Total bilirubin, Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 6 | 9
  Total bilirubin, Change from Baseline at Extension End of Treatment | -11.7758 (31.5724) | -10.6219 (24.1217)
  Direct bilirubin, Baseline of the TP: number analyzed (Participants) | 6 | 14
  Direct bilirubin, Baseline of the TP | 14.7 (2.16) | 22.9 (39.88)
  Direct bilirubin, Change from Baseline at Week 1 of the TP: number analyzed (Participants) | 5 | 8
  Direct bilirubin, Change from Baseline at Week 1 of the TP | -1.6 (4.72) | -12.1 (33.14)
  Direct bilirubin, Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 6 | 9
  Direct bilirubin, Change from Baseline at Week 2 of the TP | -0.5 (1.97) | -12.0 (33.84)
  Direct bilirubin, Change from Baseline at Week 4 of the TP: number analyzed (Participants) | 5 | 8
  Direct bilirubin, Change from Baseline at Week 4 of the TP | -1.2 (4.27) | -14.1 (38.46)
  Direct bilirubin, Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 5 | 8
  Direct bilirubin, Change from Baseline at Week 6 of the TP | -1.2 (5.89) | -14.5 (35.89)
  Direct bilirubin, Change from Baseline at Week 8 of the TP: number analyzed (Participants) | 4 | 5
  Direct bilirubin, Change from Baseline at Week 8 of the TP | 0.0 (4.24) | -22.0 (49.79)
  Direct bilirubin, Change from Baseline at Week 10 of the TP: number analyzed (Participants) | 4 | 7
  Direct bilirubin, Change from Baseline at Week 10 of the TP | -0.3 (2.99) | -13.7 (32.36)
  Direct bilirubin, Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 4 | 7
  Direct bilirubin, Change from Baseline at Week 12 of the TP | 1.0 (4.76) | -12.4 (28.98)
  Direct bilirubin, Baseline of the EP: number analyzed (Participants) | 4 | 10
  Direct bilirubin, Baseline of the EP | 14.2500 (2.6300) | 11.7000 (2.9458)
  Direct bilirubin, Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 2 | 7
  Direct bilirubin, Change from Baseline at Extension End of Treatment | -7.1322 (3.4977) | 0.1213 (6.2545)

24. Secondary Outcome: Change From Baseline in Lactate Dehydrogenase (LDH)
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Units (U)/L
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
Units (U)/L
  Baseline of the TP: number analyzed (Participants) | 10 | 14
  Baseline of the TP | 328.9 (78.34) | 469.0 (208.96)
  Change from Baseline at Week 1 of the TP: number analyzed (Participants) | 8 | 10
  Change from Baseline at Week 1 of the TP | 11.8 (70.89) | -85.1 (128.31)
  Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 9 | 11
  Change from Baseline at Week 2 of the TP | 32.2 (167.98) | -82.8 (129.32)
  Change from Baseline at Week 4 of the TP: number analyzed (Participants) | 8 | 13
  Change from Baseline at Week 4 of the TP | 65.8 (190.35) | -61.8 (152.80)
  Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 7 | 13
  Change from Baseline at Week 6 of the TP | 23.9 (133.94) | -71.4 (137.51)
  Change from Baseline at Week 8 of the TP: number analyzed (Participants) | 8 | 10
  Change from Baseline at Week 8 of the TP | 59.4 (144.20) | -66.8 (144.36)
  Change from Baseline at Week 10 of the TP: number analyzed (Participants) | 9 | 10
  Change from Baseline at Week 10 of the TP | 36.6 (118.68) | -73.5 (153.74)
  Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 8 | 13
  Change from Baseline at Week 12 of the TP | 33.8 (117.39) | -66.8 (137.28)
  Change from Baseline at Follow-up Month 2 of the TP: number analyzed (Participants) | 1 | 0
  Change from Baseline at Follow-up Month 2 of the TP | 44.0 (NA) — Standard deviation cannot be calculated for a single participant. |
  Baseline of the EP: number analyzed (Participants) | 7 | 10
  Baseline of the EP | 316.9 (86.74) | 439.8 (178.39)
  Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 5 | 8
  Change from Baseline at Extension End of Treatment | 0.0 (173.26) | 105.0 (444.64)

25. Secondary Outcome: Change From Baseline in CH50
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: microgram equivalents per Liter (µgEq/L)
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
microgram equivalents per Liter (µgEq/L)
  Baseline in the TP: number analyzed (Participants) | 9 | 14
  Baseline in the TP | 84.3 (53.91) | 69.5 (53.53)
  Change from Baseline at Week 12 in the TP: number analyzed (Participants) | 8 | 13
  Change from Baseline at Week 12 in the TP | 5.4 (21.66) | 17.2 (31.74)
  Baseline in the EP: number analyzed (Participants) | 6 | 10
  Baseline in the EP | 91.5 (52.20) | 67.6 (56.61)
  Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 1 | 1
  Change from Baseline at Extension End of Treatment | 27.0 (NA) — Standard deviation cannot be calculated for a single participant. | 12.0 (NA) — Standard deviation cannot be calculated for a single participant.

26. Secondary Outcome: Change From Baseline in Complement C3 and Complement C4
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 1638 days
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
Number analyzed (Participants) | 10 | 15
grams per Liter (g/L)
  Complement C3, Baseline of the TP: number analyzed (Participants) | 8 | 14
  Complement C3, Baseline of the TP | 0.96 (0.288) | 0.91 (0.183)
  Complement C3, Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 1 | 0
  Complement C3, Change from Baseline at Week 2 of the TP | 0.20 (NA) — Standard deviation cannot be calculated for a single participant. |
  Complement C3, Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 1 | 0
  Complement C3, Change from Baseline at Week 6 of the TP | 0.20 (NA) — Standard deviation cannot be calculated for a single participant. |
  Complement C3, Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 7 | 13
  Complement C3, Change from Baseline at Week 12 of the TP | 0.04 (0.098) | 0.12 (0.199)
  Complement C3, Baseline of the EP: number analyzed (Participants) | 5 | 10
  Complement C3, Baseline of the EP | 0.9400 (0.1949) | 0.9400 (0.1897)
  Complement C3, Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 1 | 1
  Complement C3, Change from Baseline at Extension End of Treatment | 0.1000 (NA) — Standard deviation cannot be calculated for a single participant. | 0.1400 (NA) — Standard deviation cannot be calculated for a single participant.
  Complement C4, Baseline of the TP: number analyzed (Participants) | 8 | 14
  Complement C4, Baseline of the TP | 0.1736 (0.0974) | 0.1242 (0.1046)
  Complement C4, Change from Baseline at Week 2 of the TP: number analyzed (Participants) | 1 | 0
  Complement C4, Change from Baseline at Week 2 of the TP | 0.0410 (NA) — Standard deviation cannot be calculated for a single participant. |
  Complement C4, Change from Baseline at Week 6 of the TP: number analyzed (Participants) | 1 | 0
  Complement C4, Change from Baseline at Week 6 of the TP | 0.0330 (NA) — Standard deviation cannot be calculated for a single participant. |
  Complement C4, Change from Baseline at Week 12 of the TP: number analyzed (Participants) | 7 | 13
  Complement C4, Change from Baseline at Week 12 of the TP | 0.0136 (0.0283) | 0.0274 (0.0366)
  Complement C4, Baseline of the EP: number analyzed (Participants) | 5 | 10
  Complement C4, Baseline of the EP | 0.1628 (0.0407) | 0.1160 (0.0842)
  Complement C4, Change from Baseline at Extension End of Treatment: number analyzed (Participants) | 1 | 1
  Complement C4, Change from Baseline at Extension End of Treatment | 0.0170 (NA) — Standard deviation cannot be calculated for a single participant. | 0.1100 (NA) — Standard deviation cannot be calculated for a single participant.

ADVERSE EVENTS:
Time Frame: up to a maximum of 1638 days
Description: TEAEs (adverse events either reported for the first time or the worsening of pre-existing events after the first dose of study drug) have been reported. As dose increases and decreases, based on clinical benefit and tolerability issues, respectively, were allowed during the course of the study for participants randomized to receive both 1 mg and 2.5 mg, AEs are reported per the treatment participants were randomized to rather than the dose level that was administered at the time the AE occurred.
Arm/Group | Parsaclisib 1 mg QD | Parsaclisib 2.5 mg QD
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/15
Serious Adverse Events (participants affected / at risk) | 6/10 | 5/15
Other Adverse Events (participants affected / at risk) | 10/10 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib 1 mg QD (N=10) | Parsaclisib 2.5 mg QD (N=15)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Amoebic dysentery (Infections and infestations) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Atypical mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parsaclisib 1 mg QD (N=10) | Parsaclisib 2.5 mg QD (N=15)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Asthenia (General disorders) | 1 (2) | 1 (1)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (6)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Complement factor C4 decreased (Investigations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 5 (5)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 2 (4)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lipids increased (Investigations) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 4 (4)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (7) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 2 (3)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Total complement activity decreased (Investigations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine protein/creatinine ratio increased (Investigations) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2020-11-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT03538041/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/41/NCT03538041/SAP_001.pdf